CLINICAL TRIAL: NCT00945321
Title: A Single-Dose Bioequivalence and Food Effect Study With Aprepitant and Fosaprepitant Dimeglumine in Healthy Young Adult Subjects
Brief Title: A Study to Assess the Bioequivalence of Aprepitant and Fosaprepitant and the Effect of Food on Aprepitant Bioavailability (0869-165)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0869-165; 2009_624; MK-0869-165
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Results first posted 2010-06-30 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Aprepitant; Food

ARMS (4):
- 1 (Active Comparator): aprepitant 165 mg
  Interventions: Drug: aprepitant 165 mg
- 2 (Active Comparator): aprepitant 185 mg
  Interventions: Drug: Comparator: aprepitant 185 mg
- 3 (Experimental): fosaprepitant 150 mg
  Interventions: Drug: Comparator: fosaprepitant 150 mg
- 4 (Experimental): aprepitant with food
  Interventions: Drug: Comparator: aprepitant with food

INTERVENTIONS:
Drug: aprepitant 165 mg — Single dose of aprepitant 165 mg tablet in the fasted state during treatment period 1,2, or 3.
  Arms: 1
Drug: Comparator: aprepitant 185 mg — Single dose of aprepitant 185 mg tablet in the fasted state during treatment period 1, 2, or 3.
  Arms: 2
Drug: Comparator: fosaprepitant 150 mg — Single dose of fosaprepitant 150 mg intravenous infusion in the fasted state during treatment period 1,2, or 3.
  Arms: 3
Drug: Comparator: aprepitant with food — Single dose of aprepitant 165 mg or 185 mg tablet in the fed state during treatment period 4.
  Arms: 4

SUMMARY:
This study will assess the bioequivalence of single oral doses of aprepitant (MK0869) to a single intravenous infusion of fosaprepitant (MK0517) and also determine the effect of food on the bioavailability of oral aprepitant.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Subject is a nonsmoker
* Subject is willing to comply with the study restrictions

Exclusion Criteria:

* Subject has a history of any illness that might confound the results of the study or might make participation in the study unsafe
* Subject has a history of stroke, seizures, or major neurological disorder
* Subject has a history of cancer
* Subject consumes more than two alcoholic drinks per day
* Subject consumes more than three caffeinated beverages daily

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Shadle CR, Murphy MG, Liu Y, Ho M, Tatosian D, Li SX, Blum RA. A Single-Dose Bioequivalence and Food Effect Study With Aprepitant and Fosaprepitant Dimeglumine in Healthy Young Adult Subjects. Clin Pharmacol Drug Dev. 2012 Jul;1(3):93-101. doi: 10.1177/2160763X12447304. PMID 27121336

RESULTS

PARTICIPANT FLOW:
Groups:
- A/B/C/D: Treatment A: 165 mg aprepitant Final Market Composition capsule in the fasted state/ Treatment B: 185 mg aprepitant Final Market Composition capsule in the fasted state/Treatment C: 150 mg fosaprepitant dimeglumine intravenous infusion in the fasted state/ Treatment D: 165 mg aprepitant Final Market Composition capsule in the fed state.
  (The first 12 subjects in this treatment group received a standard high-fat breakfast. The rest of the subjects (9) in this treatment group received a standard light breakfast)
- B/C/A/D: Treatment B: 185 mg aprepitant Final Market Composition capsule in the fasted state/ Treatment C: 150 mg fosaprepitant dimeglumine intravenous infusion in the fasted state/ Treatment A: 165 mg aprepitant Final Market Composition capsule in the fasted state/ Treatment D: 165 mg aprepitant Final Market Composition capsule in the fed state.
  (The first 12 subjects in this treatment group received a standard high-fat breakfast. The rest of the subjects (9) in this treatment group received a standard light breakfast)
- C/A/B/D: Treatment C: 150 mg fosaprepitant dimeglumine intravenous infusion in the fasted state/ Treatment A: 165 mg aprepitant Final Market Composition capsule in the fasted state/ Treatment B: 185 mg aprepitant Final Market Composition capsule in the fasted state/ Treatment D: 165 mg aprepitant Final Market Composition capsule in the fed state.
  (The first 12 subjects in this treatment group received a standard high-fat breakfast. The rest of the subjects (9) in this treatment group received a standard light breakfast)
- A/C/B/E: Treatment A: 165 mg aprepitant Final Market Composition capsule in the fasted state/ Treatment C: 150 mg fosaprepitant dimeglumine intravenous infusion in the fasted state/ Treatment B: 185 mg aprepitant Final Market Composition capsule in the fasted state/ Treatment E: 185 mg aprepitant Final Market Composition capsule in the fed state.
  (The first 11 subjects in this treatment group received a standard high-fat breakfast. The rest of the subjects (9) in this treatment group received a standard light breakfast)
- B/A/C/E: Treatment B: 185 mg aprepitant Final Market Composition capsule in the fasted state/ Treatment A: 165 mg aprepitant Final Market Composition capsule in the fasted state/ Treatment C: 150 mg fosaprepitant dimeglumine intravenous infusion in the fasted state/ Treatment E: 185 mg aprepitant Final Market Composition capsule in the fed state.
  (The first 11 subjects in this treatment group received a standard high-fat breakfast. The rest of the subjects (9) in this treatment group received a standard light breakfast)
- C/B/A/E: Treatment C: 150 mg fosaprepitant dimeglumine intravenous infusion in the fasted state/ Treatment B: 185 mg aprepitant Final Market Composition capsule in the fasted state/ Treatment A: 165 mg aprepitant Final Market Composition capsule in the fasted state/ Treatment E: 185 mg aprepitant Final Market Composition capsule in the fed state.
  (The first 11 subjects in this treatment group received a standard high-fat breakfast. The rest of the subjects (9) in this treatment group received a standard light breakfast)
Period: Period 1
Arm/Group | A/B/C/D | B/C/A/D | C/A/B/D | A/C/B/E | B/A/C/E | C/B/A/E
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | A/B/C/D | B/C/A/D | C/A/B/D | A/C/B/E | B/A/C/E | C/B/A/E
Started | 7 | 7 | 7 | 7 | 6 | 7
Completed | 7 | 7 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | A/B/C/D | B/C/A/D | C/A/B/D | A/C/B/E | B/A/C/E | C/B/A/E
Started | 7 | 7 | 7 | 7 | 6 | 7
Completed | 7 | 7 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | A/B/C/D | B/C/A/D | C/A/B/D | A/C/B/E | B/A/C/E | C/B/A/E
Started | 7 | 7 | 7 | 7 | 6 | 7
Completed | 7 | 7 | 7 | 7 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All randomized patients.
Arm/Group | All Participants
Number analyzed (Participants) | 42
Age, Continuous [Mean (Full Range); unit: years] | 27.8 [18 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 32
Height [Mean (Full Range); unit: Centimeters] | 172.9 [151.1 to 190.5]
Weight [Mean (Full Range); unit: Kilograms] | 74.2 [44.9 to 91.2]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC(0 to Infinity)) Following Single Dose Administration of Aprepitant 165 mg or 185 mg and Fosaprepitant 150 mg
Time Frame: Through 72 Hours Postdose
Population: All subjects excluding one subject who dropped from the study after Period 1 due to accidental overdose were included in the pharmacokinetic (PK) analysis.
Measure: Mean (Standard Deviation); unit: ng•hr/mL
Groups:
- 165 mg Aprepitant (Fasted State): 165 mg aprepitant Final Market Composition capsule in the fasted state
- 185 mg Aprepitant (Fasted State): 185 mg aprepitant Final Market Composition capsule in the fasted state
- 150 mg Fosaprepitant Dimeglumine (Fasted State): 150 mg fosaprepitant dimeglumine intravenous infusion in the fasted state
- 165 mg Aprepitant (Light): 165 mg aprepitant Final Market Composition capsule in the fed state.
  (The subjects (9) in this treatment group received a standard light breakfast.)
- 165 mg Aprepitant (High-Fat): 165 mg aprepitant Final Market Composition capsule in the fed state.
  (The (12) subjects in this treatment group received a standard high-fat breakfast.)
- 185 mg Aprepitant (Light): 185 mg aprepitant Final Market Composition capsule in the fed state.
  (The subjects (9) in this treatment group received a standard light breakfast.)
- 185 mg Aprepitant (High-Fat): 185 mg aprepitant Final Market Composition capsule in the fed state.
  (The (12) subjects in this treatment group received a standard high-fat breakfast.)
Arm/Group | 165 mg Aprepitant (Fasted State) | 185 mg Aprepitant (Fasted State) | 150 mg Fosaprepitant Dimeglumine (Fasted State) | 165 mg Aprepitant (Light) | 165 mg Aprepitant (High-Fat) | 185 mg Aprepitant (Light) | 185 mg Aprepitant (High-Fat)
Number analyzed (Participants) | 41 | 41 | 41 | 9 | 12 | 9 | 11
ng•hr/mL | 34589 (39.7) | 39053 (37.5) | 37375 (39.5) | 37795 (48.4) | 50172 (22.0) | 51146 (27.2) | 60578 (57.5)
Statistical Analysis 1: Comparison: 165 mg Aprepitant (Fasted State) vs 150 mg Fosaprepitant Dimeglumine (Fasted State); Test type: Non-Inferiority or Equivalence — Equivalence Bounds of (0.80, 1.25); p = 0.001, two one-sided tests — Hochberg's step-up procedure was applied to preserve the overall alpha level for the primary hypothesis that involved comparison at two oral dose levels; The P-value obtained was the maximum of two P-values from two one-sided tests (GMR (Oral/IV) ≤0.80 vs. GMR>0.80 and GMR≥1.25 vs. GMR<1.25); Least-Squares Mean Ratio = 0.93, 95% CI 2-sided [0.84 to 1.02]
Statistical Analysis 2: Comparison: 185 mg Aprepitant (Fasted State) vs 150 mg Fosaprepitant Dimeglumine (Fasted State); Test type: Non-Inferiority or Equivalence — Equivalence Bounds of (0.80, 1.25); p < 0.001, two one-sided tests — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least-Squares Mean Ratio = 1.05, 95% CI 2-sided [0.96 to 1.15]
Statistical Analysis 3: Comparison: 165 mg Aprepitant (Fasted State) vs 165 mg Aprepitant (High-Fat); The effect of a standard high-fat breakfast and a standard light breakfast on aprepitant plasma pharmacokinetics (AUC0-∞ and Cmax) following a single 165 mg oral dose of aprepitant and following a single 185 mg oral dose of aprepitant will be estimated in healthy young adult subjects; Test type: Superiority or Other; Least-Squares Mean Ratio = 1.47, 90% CI 2-sided [1.23 to 1.76]
Statistical Analysis 4: Comparison: 165 mg Aprepitant (Fasted State) vs 165 mg Aprepitant (Light); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Least-Squares Mean Ratio = 1.08, 90% CI 2-sided [0.88 to 1.32]
Statistical Analysis 5: Comparison: 185 mg Aprepitant (Fasted State) vs 185 mg Aprepitant (High-Fat); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Least-Squares Mean Ratio = 1.22, 90% CI 2-sided [1.01 to 1.46]
Statistical Analysis 6: Comparison: 185 mg Aprepitant (Fasted State) vs 185 mg Aprepitant (Light); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Least-Squares Mean Ratio = 1.43, 90% CI 2-sided [1.16 to 1.75]

2. Primary Outcome: Peak Plasma Concentration (Cmax) Following Single Dose Administration of Aprepitant 165 mg or 185 mg and Fosaprepitant 150 mg.
Time Frame: Through 72 Hours Postdose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | 165 mg Aprepitant (Fasted State) | 185 mg Aprepitant (Fasted State) | 165 mg Aprepitant (Light) | 165 mg Aprepitant (High-Fat) | 185 mg Aprepitant (Light) | 185 mg Aprepitant (High-Fat)
Number analyzed (Participants) | 41 | 41 | 9 | 12 | 9 | 11
ng/mL | 1738 (30.8) | 1636 (31.2) | 1870 (33.3) | 2362 (38.5) | 2116 (14.8) | 1995 (35.2)
Statistical Analysis 1: Comparison: 165 mg Aprepitant (Fasted State) vs 165 mg Aprepitant (High-Fat); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Least-Squares Mean Ratio = 1.33, 90% CI 2-sided [1.13 to 1.56]
Statistical Analysis 2: Comparison: 165 mg Aprepitant (Fasted State) vs 165 mg Aprepitant (Light); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Least-Squares Mean Ratio = 1.04, 95% CI 2-sided [0.86 to 1.25]
Statistical Analysis 3: Comparison: 185 mg Aprepitant (Fasted State) vs 185 mg Aprepitant (High-Fat); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Least-Squares Mean Ratio = 1.14, 90% CI 2-sided [0.96 to 1.34]
Statistical Analysis 4: Comparison: 185 mg Aprepitant (Fasted State) vs 185 mg Aprepitant (Light); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Least-Squares Mean Ratio = 1.40, 90% CI 2-sided [1.16 to 1.68]

ADVERSE EVENTS:
Groups:
- 165 mg Aprepitant: 165 mg aprepitant Final Market Composition capsule in the fasted state
- 185 mg Aprepitant: 185 mg aprepitant Final Market Composition capsule in the fasted state
- 150 mg Fosaprepitant Dimeglumine: 150 mg fosaprepitant dimeglumine intravenous infusion in the fasted state
- 165 mg Aprepitant (Fed State): 165 mg aprepitant Final Market Composition capsule in the fed
  state. (The first 12 subjects in this treatment group received a standard high-fat breakfast. The rest of the
  subjects (9) in this treatment group received a standard light breakfast)
- 185 mg Aprepitant (Fed State): 185 mg aprepitant Final Market Composition capsule in the fed state.
  (The first 11 subjects in this treatment group received a standard high-fat breakfast. The rest of the subjects (9) in this treatment group received a standard light breakfast)
Arm/Group | 165 mg Aprepitant | 185 mg Aprepitant | 150 mg Fosaprepitant Dimeglumine | 165 mg Aprepitant (Fed State) | 185 mg Aprepitant (Fed State)
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/42 | 0/41 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 12/41 | 13/42 | 15/41 | 6/21 | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 165 mg Aprepitant (N=41) | 185 mg Aprepitant (N=42) | 150 mg Fosaprepitant Dimeglumine (N=41) | 165 mg Aprepitant (Fed State) (N=21) | 185 mg Aprepitant (Fed State) (N=20)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 — Accidental Overdose reported for 1 subject who inadvertently received 5 capsules of 185 mg aprepitant (925 mg) instead of the protocol prescribed 1 capsule. The subject was discontinued from the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 165 mg Aprepitant (N=41) | 185 mg Aprepitant (N=42) | 150 mg Fosaprepitant Dimeglumine (N=41) | 165 mg Aprepitant (Fed State) (N=21) | 185 mg Aprepitant (Fed State) (N=20)
Eye Movement Disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chest Discomfort (General disorders) | 0 | 0 | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Infusion Site Erythema (General disorders) | 0 | 0 | 1 | 0 | 0
Infusion Site Induration (General disorders) | 0 | 1 | 2 | 0 | 0
Infusion Site Mass (General disorders) | 0 | 0 | 0 | 1 | 0
Puncture Site Indurations (General disorders) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0 | 1 | 0
Procedureal Dizziness (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 3 | 1 | 0 | 0
Headache (Nervous system disorders) | 9 | 6 | 6 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0
Oropharyngial Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Vein Pain (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.